CLINICAL TRIAL: NCT04413526
Title: The Application of Radiofrequency-assisted Liver Resection in Intractable Liver Cancer
Brief Title: Radiofrequency-assisted Liver Resection in Intractable Liver Cancer
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, head of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: radiofrequency liver resection
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Liver Cancer
Keywords: RFA; liver cancer; surgical resection
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- radiofrequency-assisted liver resection: radiofrequency-assisted liver resection for intractable liver cancer
  Interventions: Procedure: radiofrequency
- TACE(transcatheter arterial chemoembolization): temporary TACE for intractable liver cancer
  Interventions: Procedure: TACE
- radiofrequency ablation plus TACE: radiofrequency ablation plus TACE for intractable liver cancer
  Interventions: Procedure: TACE+radiofrequency

INTERVENTIONS:
Procedure: radiofrequency — radiofrequency combined with liver resection
  Groups: radiofrequency-assisted liver resection
Procedure: TACE — only TACE treatment
  Groups: TACE(transcatheter arterial chemoembolization)
Procedure: TACE+radiofrequency — TACE followed by radiofrequency
  Groups: radiofrequency ablation plus TACE

SUMMARY:
In this retrospective study, the investigators assessed the application of radiofrequency-assisted liver resection in intractable liver cancer resection, and plan to analysis the different factors.

DETAILED DESCRIPTION:
The primary clinical treatment of liver cancer is surgical resection, although many integrated applications develop rapidly, surgery is still the best way to remove the tumour lesion. Traditional ways that have curative removed tumours in three methods, which are liver resection, liver transplantation and radiofrequency ablation (RFA).

As for primary liver cancer, surgery, and RFA are both effective and safety, but for the complexity of end-stage liver cancer, surgical resection may not remove the tumours alone. Surgical resection with radiofrequency ablation therapy for intractable liver cancer is a kind of active plan. The therapy can eliminate the tumour, maximize the protection of patient liver tissue, reduce operation damage, reduce the incidence of complications, and improve patients quality of life after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound-guided fine-needle aspiration pathology or postoperative pathology was confirmed to be liver cancer, no pathological results according to China 's 2017 version of the hepatocarcinoma (HCC) diagnosis and treatment specifications, in line with the standard clinical diagnosis of liver cancer
* According to Barcelona Clinic Liver Cancer (BCLC) staging criteria, it is stage C (stage C: single tumour> 5 cm or more than three tumours, and at least one tumour> 3 cm, liver function Child-Pugh A or B, with lymph node metastasis or distant metastasis or portal vein or Venous liver trunk is invaded, penance Status (PST) score 1-2 points)

Exclusion Criteria:

* HCC patients with other malignant tumours
* Metastatic liver tumour
* Patients with liver abscess
* Patients with organ dysfunction

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCC patients
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
The survival rates for one-year to five-year | 5 years
  The survival rates was defined as the percentage of liver cancer for five years.

SECONDARY OUTCOMES:
The hospital stay | 3 months
  The length of stay in a hospital regarding days
The Child-Pugh score after therapy | 3 months
  The Child-Pugh is based on the presence and severity of ascites and hepatic encephalopathy, the prolongation of prothrombin time, and the levels of serum bilirubin and albumin. According to the Child-Pugh scores, patients are classified into three classes (Child class A, B, and C with CP scores 5-6, 7-9, and 10-15, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D., Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sun Y, Ji S, Ji H, Liu L, Li C. Clinical efficacy analysis of transcatheter arterial chemoembolization (TACE) combined with radiofrequency ablation (RFA) in primary liver cancer and recurrent liver cancer. J BUON. 2019 Jul-Aug;24(4):1402-1407. PMID 31646783